CLINICAL TRIAL: NCT03282825
Title: An Open-labelled, Parallel, Multiple Ascending Dose, Phase Ib Clinical Study of Decitabine and Paclitaxel Combination Therapy in Treating Patients With Metastatic and Locally Advanced Breast Cancer
Brief Title: Clinical Study of Decitabine and Paclitaxel Combination Therapy
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Dong Wha Pharmaceutical Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DW1018-I-1
Record Dates: First submitted 2017-09-08; First posted 2017-09-14 (Actual); Last update posted 2018-01-23 (Actual); Status verified 2018-01

CONDITIONS: Advanced Breast Cancer
MeSH Terms: interventions — Decitabine; Paclitaxel; Combined Modality Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Decitabine (Experimental): A standard 3+3 trial design will be used for Decitabine dose escalation cohorts.
  The number of cohorts is three. The subjects will be administered Decitabine on every seven days in a 28day cycle and Decitabine is sequential administered with Paclitaxel.
  Cohort 1: Decitabine 15mg/m2, Cohort 2: Decitabine 20mg/m2, Cohort 3: Decitabine 25mg/m2
  Interventions: Drug: Decitabine; Drug: Paclitaxel

INTERVENTIONS:
Drug: Decitabine — The subjects will be sequential administered with Decitabine and paclitaxel 80mg/m2 by IV(intravenous) infusion.
  Decitabine is starting dose of 15mg/m2 on 1D, 8D, 22D, 28D of a 28day cycle. Paclitaxel 80mg/m2 will be dosed in combination therapy with Decitabine on 8D, 22D, 28D of a 28day cycle.
  Other Names: DW1018
Drug: Paclitaxel — The subjects will be sequential administered with Decitabine and paclitaxel 80mg/m2 by IV(intravenous) infusion.
  Decitabine is starting dose of 15mg/m2 on 1D, 8D, 22D, 28D of a 28day cycle. Paclitaxel 80mg/m2 will be dosed in combination therapy with Decitabine on 8D, 22D, 28D of a 28day cycle.
  Other Names: combination therapy

SUMMARY:
Phase Ib clinical study of Decitabine and Paclitaxel combination therapy

DETAILED DESCRIPTION:
An open-labelled, parallel, multiple ascending dose, phase Ib clinical study of Decitabine and Paclitaxel combination therapy in treating patients with metastatic and locally advanced breast cancer

ELIGIBILITY:
Inclusion Criteria:

1. age ≥ 19 years as female
2. be unable to operate for therapy with HER2 negative breast adenocarcinoma and metastatic breast cancer, one or more chemotherapy
3. according to RECIST ver.1.1, one or more evaluable lesion
4. Eastern cooperative oncology group(ECOG) performance score is o or 1
5. lesion for core biopsy
6. Within 28days of planned first study treatment day, laboratory safety test is satisfied. ANC ≥1500cells/microliter, Platelet count ≥ 100,000 cells/microliter, Hemoglobin≥8.5g/dl, ALT and AST ≤ 2ULN, ALP≤2.5ULN, Serum total bilirubin≤1.25 ULN, PT-INR and aPTT≤1.5ULN, Creatinine≥50ml/min
7. menopause or informed that effective contraception must be used during the entire treatment period of this study and for 6 months after exiting from the study
8. Given signed and dated written informed consent form

Exclusion Criteria:

1. Symptomatic metastasis and Leptomeningeal metastasis
2. Injection of paclitaxel for metastatic breast cancer within 6 months
3. HER2, Positive Breast adenocarcinoma
4. cancertherapy for whole body within 3 weeks
5. radiotherapy for metastatic region within 4 weeks
6. major surgery, open biopsy and trauma within 4 weeks
7. less than 4 weeks post major surgery
8. treatment with consistently systemic corticosteroid or immunosuppressive drug
9. more than 2 grade for peripheral neuropathy
10. Congenital ling QT syndrome or QTc interval > 480 milisecond
11. occur myocardial infartion within 6 months
12. unstable angina pectoris
13. HIV(+) or AIDS
14. HBsAg(+) or HCV(+)
15. treatment bisphosphonate for hypercalcemia
16. except metastatic and locally advanced breast cancer, personal history with malignancy within 5 years
17. hypersensitivity reaction with paclitaxel or Cremophor EL formulation
18. Pregnant or breast feeding
19. be unable or unwilling to abide by the study protocol or to cooperate fully with the investigator or designee

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2017-03-28 (Actual); Primary Completion 2018-02 (Estimated); Study Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerant Dose (MTD) and Dose Limiting Toxicity (DLT) | for about 4 weeks
  According to principle of Dose Limited Toxicity (DLT) assessment by National Cancer Institute Common Terminonlgy Criteria for Adverse Events (NCI-CTCAE, V4.0), DLT is evaluated above grade 3 as adverse event.

CONTACTS AND LOCATIONS:
Overall Officials: Joo Hyuk Sohn, MD, PhD, Principal Investigator — Yonsei University Health System, Severance Hospital
Locations (1):
- Yonsei University Health System, Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No